CLINICAL TRIAL: NCT00645944
Title: Randomized, Controlled, Double Blind Trial of Eszopiclone for Insomnia Associated With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Cenk Tek, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0702002331; ESRC131
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Insomnia; Schizophrenia; Schizoaffective Disorder; Sleep Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Schizophrenia; Psychotic Disorders; Sleep Wake Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone Group (Experimental): Participants assigned to this arm will receive Eszopiclone 2mg each night for the first week then Eszopiclone 3mg each night for the remaining weeks.
  Interventions: Drug: Eszopiclone
- Placebo Group (Placebo Comparator): Participants assigned to this arm will receive placebo (an inactive substance or a "sugar pill") to be taken each night for all weeks of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 2mg each night for the first week then Eszopiclone 3mg each night for the remaining weeks.
  Other Names: Lunesta
  Arms: Eszopiclone Group
Drug: Placebo — Placebo or inactive substance ("sugar pill")taken each night for all weeks of the study
  Arms: Placebo Group

SUMMARY:
The major goal of this project is to investigate established insomnia treatments in a schizophrenia population to see if the improved sleep leads to overall better quality of life. In addition, we hypothesize that the insomnia treatment may also lead to observed improvements in other symptoms associated with schizophrenia such as cognitive impairments, obesity, and negative symptoms.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the clinical efficacy of eszopiclone for the treatment of schizophrenia-related insomnia over 8 weeks. A two-week, single-blind placebo phase followed the double-blind phase to evaluate rebound and withdrawal effects after abrupt discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 to 64
* Meet DSM-IV criteria for schizophrenia or schizoaffective disorder
* Sleep difficulties at least 2x per week in the preceding month
* Be on a stable dose of antipsychotic medication
* Symptomatically stable in the last 2 months
* English speaking.

Exclusion Criteria:

* Meet criteria for current alcohol or other substance dependence
* A history of dementia, mental retardation or other neurological disorder
* Not capable of giving informed consent for participation in this study.
* Ongoing pregnancy
* Known sensitivity to zopiclone.
* Insomnia associated with medical disorders likely to impair sleep.
* Use of any medication that affects sleep/wake function (other than antipsychotic medication), within the past 2 weeks or within a time period that is less than 7 half-lives since last use of the medication.
* Lack of sleep benefit from previous adequate eszopiclone treatment
* History of clinically significant hepatic impairment.
* Subject is taking a potent cytochrome p450 3A4 inhibitor medication (ritonavir, nelfinavir, indinavir, erythromycin, clarithromycin, troleandomycin, ketoconazole, itraconazole) and is unwilling or it is clinically contraindicated to stop the medication.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between May 2008 and February 2011 at a community mental health center. Following screening and baseline assessment, eligible patients who continued to meet inclusion criteria were randomly assigned to either placebo or eszopiclone in a 1:1 ratio using a randomization procedure blind to both research team and subjects.
Pre-assignment Details: 179 outpatients were screened, 44 met initial eligibility criteria. Forty-three consented to participate and 4 were withdrawn prior to randomization. Of the remaining 39, 19 were randomized to placebo and 20 to eszopiclone 3mg. Two participants in the placebo arm and 1 participant in the eszopiclone arm withdrew before receiving study medication
Period: Randomized
Arm/Group | Eszopiclone Group | Placebo Group
Started | 20 | 19
Completed | 19 | 17
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Received Medication
Arm/Group | Eszopiclone Group | Placebo Group
Started | 19 | 17
Completed | 13 | 14
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the remaining 39 randomized, 19 were randomized to placebo and 20 to eszopiclone 3mg. Two participants in the placebo arm and 1 participant in the eszopiclone arm withdrew before receiving study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone Group | Placebo Group | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (7.4) | 47.5 (10.2) | 46.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index From Baseline.
Description: The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire that provides a global measure of insomnia severity based on several indicators (e.g., difficulty falling or staying asleep, satisfaction with sleep, degree of impairment with daytime functioning). It has adequate internal consistency (Cronbach's alpha=0.91) and temporal stability (r=0.80), has been validated against sleep diary and polysomnography data and was sensitive to change in several insomnia treatment studies. The ISI scale range is: minimum = 0, maximum = 28. The interpretation is that lower is 'better sleep', while higher is considered 'worse sleep/more insomnia'.
Time Frame: 8 Weeks
Population: Of 39 eligible participants, 19 were randomized to placebo and 20 to eszopiclone 3mg. Two participants in the placebo arm and 1 participant in the eszopiclone arm withdrew before receiving study medication. 36 participants were included in the modified ITT analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Eszopiclone Group | Placebo Group
Number analyzed (Participants) | 19 | 17
units on a scale | -10.7 [-13.2 to -8.2] | -6.9 [-9.5 to -4.3]
Statistical Analysis 1: Comparison: Eszopiclone Group vs Placebo Group; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-7.5 to -0.2]

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Adverse events reported in either placebo or eszopiclone group during double blind phase at 8 weeks.
Arm/Group | Eszopiclone Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 3/19 | 1/17
Other Adverse Events (participants affected / at risk) | 16/19 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone Group (N=19) | Placebo Group (N=17)
Unpleasant Taste (General disorders) | 1 (1) | 1 (1) — Participants dropped out of the study due to the unpleasant taste of the intervention/placebo.
Fatigue (General disorders) | 1 (1) | 0 (0)
Memory Problems (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone Group (N=19) | Placebo Group (N=17)
Sedation/drowsiness (General disorders) | 8 (8) | 7 (7)
Fatigue/Weakness (General disorders) | 2 (2) | 1 (1)
Irritability (General disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Excitement/nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Malaise (Psychiatric disorders) | 3 (3) | 0 (0)
Memory Problems (Nervous system disorders) | 0 (0) | 1 (1)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness/faintness (Nervous system disorders) | 2 (2) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dry Mouth (General disorders) | 5 (5) | 4 (4)
Increased Salivation (General disorders) | 1 (1) | 1 (1)
Unpleasant Taste (General disorders) | 7 (7) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) — Ataxia/impaired coordination
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomach/ abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urination Problems (Renal and urinary disorders) | 0 (0) | 1 (1)
Libido Decrease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Orgasmic Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Sweating excessively
Appetite Decrease (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Appetite Increase (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Other (General disorders) | 1 (1) | 3 (3) — Other unspecified non-serious adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No